CLINICAL TRIAL: NCT02475876
Title: Pharmacokinetics of Clindamycin and Trimethoprim-sulfamethoxazole in Infants and Children Using PBPK
Brief Title: PK of Clindamycin and Trimethoprim-sulfamethoxazole in Infants and Children
Acronym: PBPK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Cohen-Wolkowiez (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Michael Cohen-Wolkowiez, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00057185; 1R01HD076676-01A1 (NIH)
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Clindamycin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- clindamycin (Other): Each subject will be assigned to study drug (clindamycin or TMP-SMX) at the discretion of the treating clinician. The dose and dosing interval of study drug are dictated by this protocol (see interventions).
  Interventions: Drug: Clindamycin
- trimethoprim-sulfamethoxazole (Other): Each subject will be assigned to study drug (clindamycin or TMP-SMX) at the discretion of the treating clinician. The dose and dosing interval of study drug are dictated by this protocol (see interventions).
  Interventions: Drug: trimethoprim-sulfamethoxazole

INTERVENTIONS:
Drug: Clindamycin — Route of administration is IV for all Cohorts. Dosing interval is every 8 hrs. for all Cohorts:
  * Cohort 1; No. Subjects = 5; Age 1-5 months; Dose = 9 mg/kg;
  * Cohort 2; No. Subjects = 5; Age >5 months to 1 year; Dose =12 mg/kg;
  * Cohort 3; No. Subjects = 5; Age >1-2 years; Dose =12 mg/kg.
  * Cohort 4; No. Subjects = 4; Age >2-6 years; Dose =12 mg/kg.
  * Cohort 5; No. Subjects = 4; Age >6-12 years; Dose =10 mg/kg.
  * Cohort 6; No. Subjects = 4; Age >12-16 years; Dose =10 mg/kg.
  Other Names: Cleocin
  Arms: clindamycin
Drug: trimethoprim-sulfamethoxazole — Route of administration is PO for all Cohorts. Dosing interval is every 12 hrs. for all Cohorts:
  * Cohort 1; No. Subjects = 5; Age 1-5 months; Dose = 6 mg/kg.
  * Cohort 2; No. Subjects = 5; Age >5 months to 1 year; Dose = 6 mg/kg.
  * Cohort 3; No. Subjects = 5; Age >1-2 years; Dose = 6 mg/kg.
  * Cohort 4; No. Subjects = 4; Age >2-6 years; Dose = 6 mg/kg.
  * Cohort 5; No. Subjects = 4; Age >6-12 years; Dose = 6 mg/kg.
  * Cohort 6; No. Subjects = 4; Age >12-16 years; Dose = 4 mg/kg.
  Other Names: Bactrim, TMP-SMX
  Arms: trimethoprim-sulfamethoxazole

SUMMARY:
Developmental changes in physiology during childhood influence drug dosing. Failure to account for these changes leads to improper dosing, which is associated with decreased drug efficacy and safety in children. Population physiologically-based pharmacokinetic (PBPK) modeling offers the opportunity to predict optimal drug dosing based on physiologic parameters adjusted for developmental changes.

PBPK models are mathematical constructs that incorporate physiologic processes with drug characteristics and genetic variances to characterize the dose-exposure relationship across the age continuum. These models integrate drug-specific (e.g., metabolism, protein binding) and systems-specific (e.g., organ size, blood flow) information to predict the effect of different factors (e.g., age, genetic variants, disease) on drug exposure. By accounting for these factors and using data from clinical trials to confirm the modeling, PBPK models can reduce the number of children needed for clinical trials while maximizing dose-based efficacy and safety.

This trial will evaluate a platform to prospectively validate population PBPK models in children. The study drugs, clindamycin and Bactrim (aka TMP-SMX), are ideal candidates to evaluate population PBPK models in children due to their differing physico-chemical properties and elimination pathways. In addition, a trial of clindamycin and TMP-SMX has broad clinical applicability, as both drugs are among the most commonly used agents to treat gram-positive infections in infants and children.

DETAILED DESCRIPTION:
This is a PK and safety study in infants and children requiring prophylaxis of, or treatment for confirmed or suspected infection with clindamycin or TMP-SMX. Each subject will be involved in the study for up to 33 days (3 days of therapy, 30 days for serious adverse event monitoring).

STUDY PROCEDURES

Baseline/pre-dose assessment - After the parent or legally authorized representative has signed the IRB-approved informed consent form and after it has been determined that the subject satisfies all inclusion and no exclusion criteria, the following evaluations will be recorded in the CRF:

1. Subject demographics including sex, date of birth, race, and ethnicity
2. For infants ≤12 months of age: gestational age (GA) and body weight at birth
3. Active medical history (from admission note in medical record)
4. Concomitant medications
5. For subjects receiving study drugs per standard of care, record the last 6 doses of clindamycin or TMP-SMX received prior to study drug administration (date, time, route of administration)
6. Targeted physical examination, including weight and length/height
7. Laboratory determinations within 48 hours prior to enrollment if performed per local standard of care. If serum creatinine was not collected as standard of care, it will be collected for this study to confirm eligibility.
8. Microbiology determinations within 48 hours prior to enrollment if performed per local standard of care.

Treatment assessments/procedures (Day 1-3) - The following assessments will be conducted each day while the subject is on study:

1. Date, time, route, site of administration, dose, and formulation of each study drug dose
2. Concomitant medications
3. PK sampling (blood and urine) with date, time, and site of collection
4. Genetic sampling (once)
5. Laboratory determinations if performed per standard of care
6. Microbiologic determinations if performed per standard of care
7. Serum sample for determination of alpha-1-acid glycoprotein concentration for subjects enrolled in the clindamycin arm only. Alpha-1-acid glycoprotein concentration will be measured in one of the plasma PK samples. A separate blood sample is not required.
8. Study drug-related adverse events AEs and SAEs If available, record laboratory determinations daily; if several laboratory determinations are available for the same day, record test results closest to administration of study drug.

PK SAMPLING

Plasma pharmacokinetics sampling scheme.

Clindamycin: Sample collection windows are relative to the start of the infusion for IV clindamycin, except for the first post-infusion sample, which is relative to the end of the infusion.

Three plasma PK samples will be collected around the first dose according to the following sampling windows:

* 0-10 minutes after the end of the first dose
* 2-4 hours after the start of the first dose
* <30 minutes prior to second dose

Four plasma PK samples will be collected any time after dose 6 according to the following sampling windows.

* Pre-dose
* 0-10 minutes
* 2-4 hours
* <30 minutes prior to next scheduled dose

While treatment with IV clindamycin is necessary for inclusion in the clindamycin arm of the study, subjects may transition from IV to oral clindamycin and be eligible for PK sample collection during the oral phase.

TMP-SMX: Sample collection windows are relative to the administration of oral TMP-SMX.

Three plasma PK samples will be collected around the first dose according to the following sampling windows:

* 1-3 hours after the end of the first dose
* 6-8 hours after the start of the first dose
* <30 minutes prior to second dose

Four plasma PK samples will be collected any time after dose 6 according to the following sampling windows.

* Pre-dose
* 1-3 hours
* 6-8 hours
* <30 minutes prior to next scheduled dose

Urine PK samples - Urine PK samples are not required for a subject to complete the study. If possible, every effort should be made to collect urine PK samples according to the following schedule.

Clindamycin IV: One urine sample will be collected as timed aliquots of all urine excreted during one of the following intervals after dose 6:

* 0-2 hours
* 2-4 hours
* 4-8 hours

TMP-SMX: One urine sample will be collected as timed aliquots of all urine excreted during one of the following intervals after dose 6:

* 0-3 hours
* 3-6 hours
* 6-9 hours
* 9-12 hours

Opportunistic PK samples - Opportunistic samples of bone, skin, and synovial fluid will also be collected if obtained per standard of care.

Sampling for genotyping - All blood pellets left over after centrifugation of each plasma PK samples will be collected and combined into one whole blood pellet sample per subject. This combined whole blood pellet will be sent for genetic analysis of single nucleotide polymorphisms in the CYP3A family and CYP2C9 genes.

STATISTICS

All subjects who receive at least 1 dose of study drug will be included in the intention-to-treat (ITT) population used for the safety analysis. All subjects who provide at least 1 evaluable PK sample will be included in the PK analysis. Descriptive statistics such as number of observations, mean, median, standard deviation, standard error, minimum, and maximum will be presented for continuous variables (such as age, weight, etc.). Other descriptive statistics such as counts, proportions, and/or percentages will be presented to summarize discrete variables (such as race, sex, etc.). All descriptive analyses will be presented by appropriate treatment group (ITT or per-protocol) and overall. A detailed description of statistical methods and secondary analyses will be prepared and presented in the statistical analysis plan prior to data lock for final analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from parent or guardian and assent from subject when appropriate
2. Require prevention or treatment of confirmed or suspected infection
3. PMA >36 weeks
4. Able to take oral drugs (TMP-SMX)
5. Sufficient IV access for study drug administration (for clindamycin) and PK sample collection (both drugs) -

Exclusion Criteria:

1. History of allergic reactions to study drugs
2. Treatment with the following drugs within 24 hours prior to first dose of clindamycin or expected to receive these drugs during the treatment phase with clindamycin:

   * CYP3A4 inhibitors (nefazodone, fluconazole, ketoconazole, fluvoxamine, conivaptan, diltiazem, verapamil, aprepitant, ticlopidine, crizotinib, and imatinib), or
   * CYP3A4 inducers (rifampin, phenytoin, carbamazepine, phenobarbital, troglitazone, pioglitazone, and St. John's wort).
3. Serum creatinine >2 mg/dl within 48 hours prior to enrollment
4. Known ALT >250 U/L or AST >500 U/L on measurement closest to the time of enrollment
5. Known pregnancy
6. Breastfeeding females
7. On extracorporeal membrane oxygenation support at the time of study drug dosing or PK sampling
8. Any condition that, in the judgment of the investigator, precludes participation because it could affect subject safety -

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2015-11; Primary Completion 2018-08-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration at steady state (Cmaxss) - clindamycin | PK sampling taken during 3 continuous days of treatment
  We will use the population PBPK models to simulate drug concentration vs. time data for each individual subject using the characteristics and genetic information of the subjects enrolled in the study. We will compare simulated vs. observed plasma concentrations.
Area under the plasma concentration versus time curve from the start to the end of one dosing interval at steady state (AUCss) - clindamycin | PK sampling taken during 3 continuous days of treatment
  We will use the population PBPK models to simulate drug concentration vs. time data for each individual subject using the characteristics and genetic information of the subjects enrolled in the study. We will compare simulated vs. observed plasma concentrations.
Maximum observed plasma concentration at steady state (Cmaxss) - Trimethoprim-Sulfamethoxazole | PK sampling taken during 3 continuous days of treatment
  We will use the population PBPK models to simulate drug concentration vs. time data for each individual subject using the characteristics and genetic information of the subjects enrolled in the study. We will compare simulated vs. observed plasma concentrations.
Area under the plasma concentration versus time curve from the start to the end of one dosing interval at steady state (AUCss) - Trimethoprim-Sulfamethoxazole | PK sampling taken during 3 continuous days of treatment
  We will use the population PBPK models to simulate drug concentration vs. time data for each individual subject using the characteristics and genetic information of the subjects enrolled in the study. We will compare simulated vs. observed plasma concentrations.

SECONDARY OUTCOMES:
Number of reported AEs and SAEs | 33 days
  Number of AEs and SAEs reported during (3 continuous days) and up to 30 days after study drug administration
Number of Subjects Heterozygous for any CYP3A Family Genotype | 33 days
  Genetic analysis of the most important single nucleotide polymorphisms (SNPs) in the CYP3A family and CYP2C9 genes will be performed using commercially available Taqman Polymerase Chain Reactions assays for the following gene expressions:
  CYP3A4: rs35599367, rs2246709, rs4646437, rs2740565, rs4253728 CYP3A5: rs776746, rs10264272, rs15524 CYP3A7: rs2687133, rs2257401 CYP2C9: rs1799853, rs1057910
  Subjects will be classified into homozygous and heterozygotes for allelic variants based on the genotyping results.
Number of Subjects Heterozygous for any CYP2C9 Genotype | 33 days
  Genetic analysis of the most important single nucleotide polymorphisms (SNPs) in the CYP3A family and CYP2C9 genes will be performed using commercially available Taqman Polymerase Chain Reactions assays for the following gene expressions:
  CYP3A4: rs35599367, rs2246709, rs4646437, rs2740565, rs4253728 CYP3A5: rs776746, rs10264272, rs15524 CYP3A7: rs2687133, rs2257401 CYP2C9: rs1799853, rs1057910
  Subjects will be classified into homozygous and heterozygotes for allelic variants based on the genotyping results.
Number of Subjects Homozygous for any CYP3A Family Genotype | 33 days
  Genetic analysis of the most important single nucleotide polymorphisms (SNPs) in the CYP3A family and CYP2C9 genes will be performed using commercially available Taqman Polymerase Chain Reactions assays for the following gene expressions:
  CYP3A4: rs35599367, rs2246709, rs4646437, rs2740565, rs4253728 CYP3A5: rs776746, rs10264272, rs15524 CYP3A7: rs2687133, rs2257401 CYP2C9: rs1799853, rs1057910
  Subjects will be classified into homozygous and heterozygotes for allelic variants based on the genotyping results.
Number of Subjects Homozygous for any CYP2C9 Genotype | 33 days
  Genetic analysis of the most important single nucleotide polymorphisms (SNPs) in the CYP3A family and CYP2C9 genes will be performed using commercially available Taqman Polymerase Chain Reactions assays for the following gene expressions:
  CYP3A4: rs35599367, rs2246709, rs4646437, rs2740565, rs4253728 CYP3A5: rs776746, rs10264272, rs15524 CYP3A7: rs2687133, rs2257401 CYP2C9: rs1799853, rs1057910
  Subjects will be classified into homozygous and heterozygotes for allelic variants based on the genotyping results.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cohen-Wolkowiez, MD, Principal Investigator — Duke Clinical Research Institute
Locations (3):
- United States (3):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan

REFERENCES:
- [Derived] Wu YSS, Cohen-Wolkowiez M, Hornik CP, Gerhart JG, Autmizguine J, Cobbaert M, Gonzalez D; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. External Evaluation of Two Pediatric Population Pharmacokinetics Models of Oral Trimethoprim and Sulfamethoxazole. Antimicrob Agents Chemother. 2021 Jun 17;65(7):e0214920. doi: 10.1128/AAC.02149-20. Epub 2021 Jun 17. PMID 33903114